CLINICAL TRIAL: NCT07243197
Title: Safety and Performance Evaluation Study of DragonFly M2 System for Mitral Regurgitation
Brief Title: DragonFly M2 Pivotal Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hangzhou Valgen Medtech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DragonFly-M2 01
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Mitral Valve (MV) Regurgitation
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DragonFly M2 Transcatheter Mitral Valve Repair System (Experimental): Transcatheter mitral valve repair with the DragonFly M2 System in patients with degenerative mitral regurgitation
  Interventions: Device: DragonFly M2 Transcatheter Mitral Valve Repair System

INTERVENTIONS:
Device: DragonFly M2 Transcatheter Mitral Valve Repair System — Edge-to-edge repair with DragonFly M2 System

SUMMARY:
To confirm the effectiveness and safety of the DragonFly M2 Transcatheter Mitral Valve Repair System for the treatment of symptomatic moderate-to-severe (3+) or severe (4+) degenerative mitral regurgitation in high surgical risk subjects.The safety and effectiveness of the first-generation device(Dragonfly Transcatheter Mitral Valve Repair System)have been previously demonstrated. This study aims to further confirm the safety and effectiveness of the new device following structural optimization based on the first-generation design.

DETAILED DESCRIPTION:
This is a prospective, multicentric clinical investigation.

Subjects to be included in this clinical investigation suffer from symptomatic chronic moderate-to-severe (3+) or severe (4+) DMR with high or prohibitive surgical risk judged by a local investigation site's heart team .

After signing an informed consent form, subjects in the experimental group will undergo the transcatheter mitral valve repair procedure using the DragonFly M2 Transcatheter Mitral Valve Clip System. All subjects were followed up immediately after procedure, before discharge, 30 days , 6 months, 12 months after procedure, and 2, 3, 4, and 5 years after procedure.

ELIGIBILITY:
Inclusion Criteria:

1.≥ 18 years old. 2.Moderate to severe (3+) or severe (4+) chronic DMR determined by transthoracic echocardiography.

* Transseptal catheterization is determined to be feasible by the Investigator.
* Patients have been informed of the nature of the study, understand the purpose of the clinical trial, voluntarily participate in the study, and sign the ICF.

Exclusion Criteria:

1)Echocardiographic evidence of intracardiac mass, thrombus, or vegetation. 2) The presence of other severe heart valve disease requiring surgical intervention.

3) Prior mitral valve leaflet surgery or transcatheter mitral valve intervention.

* Currently participating in an investigational drug or another device study that has not completed its primary endpoints or would clinically interfere with the endpoint of this study. Note: Trials requiring extended follow-up for products that were investigational, but have since become commercially available, are not considered investigational trials.
* In the judgment of the investigator, subjects may not complete the trial according to poor compliance or in other circumstances when the investigator determines that the subject is unfit to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2031-06-30 (Estimated)

PRIMARY OUTCOMES:
Procedure success | 30 Days
  Procedure success: device implanted successfully, MR ≤ 2+ at discharge (or 30-day echo if unavailable), and no death or device-related reintervention within 30 days post-procedure.

SECONDARY OUTCOMES:
Single-click release success | Intraoperative
  successful clip detachment from the delivery system at the intended position during the first release attempt
Acute device success | Immediately after procedure
  One or more Dragonfly devices are successfully delivered and released, edge-to-edge leaflet repair confirmed by echocardiogram, and successfully withdrawal of the delivery catheter.
surgical intervention | 30 days, 6 months, and 12 months
  surgical interventions due to post-procedural mitral valve dysfunction
NYHA Class | 30 days, 6 months, and 12 months
  Number of patients with New York Heart Association (NYHA) Function Class I or II.
Quality of life improvement | 30 days, 6 months, and 12 months
  Improvement in quality of life (QoL) over baseline, as measured by the Kansas City Cardiomyopathy Questionnaire (KCCQ).

OTHER OUTCOMES:
Incidence of major adverse events (MAEs) | 30 days, 6 months, and 12 months
  MAE is defined as a combined clinical endpoint of death, stroke, myocardial infarction, renal failure, and nonelective cardiovascular surgery for device or procedure-related adverse events occurring after transseptal catheterization.
All-cause mortality | 30 days, 6 months, and 12 months
  Percentage of all-cause death includes cardiac death, non-cardiac death, and death from unknown causes.
Cardiovascular death | 30 Days, 6 months, 12 months
  Cardiovascular death

CONTACTS AND LOCATIONS:
Overall Officials: Xiangbin Pan, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Fuwai Hospital Chinese Academy of Medical Sciences, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No